CLINICAL TRIAL: NCT02887560
Title: Comparison by Transoesophageal Assessement of Systolic Right Ventricle Function Measures in Perioperative Care of Pulmonary Transplant.
Acronym: ETO VD PERIOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 6283
Record Dates: First submitted 2016-06-20; First posted 2016-09-02 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Primary Lung Graft Dysfunction
Keywords: Right ventricle; Pulmonary transplantation; Strain; isovolumic acceleration (IVA)
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patient (Experimental): Only one arm has been specified for the protocol. This arm included all study patient (33) for which the intervention is to be administered
  Interventions: Procedure: transoesophageal echocardiography

INTERVENTIONS:
Procedure: transoesophageal echocardiography

SUMMARY:
The aim of the study is to describe the early adaptation of the right ventricle assessed by echocardiography to change of pulmonary circulation secondary to pulmonary transplantation.

Secondary objectives include change of haemodynamics measured by transpulmonary thermodilution and evolution of right heart function in terms of primary graft dysfunction grading.

ELIGIBILITY:
Inclusion Criteria:

* Adult (over 18 years)
* Patient affiliated to a social protection scheme insurance
* Patient was informed of the study and w gave their consent
* Patient on the lung transplant list
* Patient eligible for a pulmonary transplantation after decision of a multidisciplinary team
* Patients with chronic lung disease with parenchymal dysfunctions (Chronic obstructive pulmonary disease or COPD, alpha-1 antitrypsin deficiency, cystic fibrosis, pulmonary fibrosis, bronchiolitis obliterans organizing pneumonia or BOOP)

Exclusion Criteria:d

* Minor patients
* Patient under judicial protection, under guardianship
* Patient in exclusion period (determined by a previous study or in progress)
* Patient participating in parallel in another clinical trial that may interfere with the results of the study
* Inability to give informed patient information (emergency, understanding difficulties, etc ...)
* The refusal of patient consent
* The use of cardiopulmonary bypass during lung transplantation
* Uni-pulmonary transplant
* A transplant for idiopathic or primary pulmonary hypertension
* The presence of a cons-indication for transesophageal echocardiography:

  o Absolute contraindications:
* Abnormalities of the esophagus: stenosis, tumor, diverticulum perforation, active bleeding

  o Relative contraindications:
* ancient cervicothoracic irradiation history (> 10 years)
* recent upper gastrointestinal bleeding history
* presence of esophageal varices ≥ grade II
* zero cervical mobility
* Reflux Esophagitis
* Severe coagulation disorders
* Pregnancy / Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-27 (Actual)

PRIMARY OUTCOMES:
Transesophageal echocardiographic assessment for comparision of right ventricle free-wall strain rate in perioperative care of bipulmonary transplantation | Outcome is measured 3 times : after induction of general anesthesia, before surgical incision, after throacic closure and 6 to 12 hours postoperative.
Transesophageal echocardiographic assessment for comparision of right ventricle isovolumic acceleration in perioperative care of bipulmonary transplantation | utcome is measured 3 times : after induction of general anesthesia, before surgical incision, after throacic closure and 6 to 12 hours postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Gharib Ajob, MD, Principal Investigator — Strasbourg's University Hospitals
Locations (1):
- Strasbourg's New Civil Hospital, Cardiac surgical reanimation department, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No